CLINICAL TRIAL: NCT00642434
Title: Carvedilol vs.Metoprolol: A Comparison of Effects on Endothelial Function and Oxidative Stress in Response to Acute Hyperglycemia in Patients With Type 2 Diabetes and Hypertension
Brief Title: Comparison of Blood Pressure Medications on Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: UNM04094
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
Keywords: diabetes blood pressure oxidative stress
MeSH Terms: conditions — Diabetes Mellitus | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): study drug- carvedilol
  Interventions: Drug: carvedilol
- 2 (Active Comparator): study drug metorprolol
  Interventions: Drug: metoprolol

INTERVENTIONS:
Drug: carvedilol — variable
  Other Names: coreg; toprol
  Arms: 1
Drug: metoprolol — variable
  Arms: 2

SUMMARY:
The purpose of this study is to determine if there are differences, (benefits) between carvedilol and metoprolol in the treatment of HTN in patients with type 2 diabetes. Specifically we will be looking at differences in blood pressure and blood sugar control, endothelial function, inflammation, oxidative stress and coagulation.

Subjects will be randomized to one of the two beta-blockers and followed for 5 months. Each subject will undergo 4 inpatient studies where an oral glucose tolerance test will be done, Inflammatory and oxidative stress markers will be measured. Endothelial function will be measured using brachial artery ultrasound and laser skin Doppler

DETAILED DESCRIPTION:
The purpose of this study is to determine if there are differences, (benefits) between carvedilol and metoprolol in the treatment of HTN in patients with type 2 diabetes. Specifically we will be looking at differences in blood pressure and blood sugar control, endothelial function, inflammation, oxidative stress and coagulation.

Subjects will be randomized to one of the two beta-blockers and followed for 5 months. Each subject will undergo 4 inpatient studies where an oral glucose tolerance test will be done, Inflammatory and oxidative stress markers will be measured. Endothelial function will be measured using brachial artery ultrasound and laser skin Doppler. Baseline visit will be done when subjects are off all antihypertension medications except ACEI/ARB. Following the baseline study subjects will be randomized to study drug. The dose will be titrated until goal blood pressure is reached. Add on medication will be used if needed.

Subjects will then undergo a second study. The third study will take place after 5 months on treatment. Stud drug will then be stoppped and subjects will be restudied 2 weeks later

ELIGIBILITY:
Inclusion Criteria:

* not enrolling

Exclusion Criteria:

* not enrolling

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UNMHSC, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Colleran K, Aguirre L, Burge MR. Carvedilol vs. metoprolol: A comparison of effects on endothelial function and oxidative stress in response to acute hyperglycemia in patients with type 2 diabetes and hypertension. Journal of Diabetes Mellitus 2(1):146-151, 2012.

RESULTS

PARTICIPANT FLOW:
Groups:
- Metoprolol: Randomized to Metoprolol
- Carvedilol: Radomized to Carvedilol
Period: Overall Study
Arm/Group | Metoprolol | Carvedilol
Started | 10 | 12
Number of Participants Treated | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Number of Participants Treated With Metoprolol: Randomized to Metoprolol
- Number of Participants Treated With Carvedilol: Radomized to Carvedilol
- Total: Total of all reporting groups
Arm/Group | Number of Participants Treated With Metoprolol | Number of Participants Treated With Carvedilol | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were not collected

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Change in Markers of Inflammation (PAI-1) Following Treatment Compared to Baseline
Description: Reporting the number of participants with a change in markers of inflammation (PAI-1) following treatment compared to baseline.
Time Frame: 5 months
Measure: Number; unit: participants
Arm/Group | Metoprolol | Carvedilol
Number analyzed (Participants) | 9 | 11
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: PI left institution and study withdrawn.
Description: PI left institution and study withdrawn.
Arm/Group | Metoprolol | Carvedilol
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes